CLINICAL TRIAL: NCT03014518
Title: Peripheral Neuroinflammatory Predictors of Suicidal Risk at Time of Inpatient Discharge in Adolescents
Brief Title: Biomarkers as Predictors of Suicidal Risk in Adolescents
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Case Western Reserve University (Other); Van Andel Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tatiana Falcone, MD, Staff, Cleveland Clinic, The Cleveland Clinic
Other Study IDs: 16-630; MH108857 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2016-12-15; First posted 2017-01-09 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Suicide, Attempted; Suicidal Ideation; Suicidal Intention; Suicide
Keywords: Adolescent; Biological Markers; Biomarkers; Biomarkers for suicidality; Blood brain barrier; Clinical predictors; Cytokine; Feeling suicidal; Inflammation; Inflammatory marker; Inpatient discharge; Interleukin-1 beta; IL-1ß; Interleukin-6; IL-6; Kynurenic acid; Kynurenine pathway; Neuroinflammation; Novel marker; Peripheral blood biomarkers; Picolinic acid; Plasma biomarker; Psychiatric inpatient; S100B; Serum biomarker; Stress; Suicide; Suicidal behavior; Suicidal risk; Tumor necrosis factor alpha; TNF-α
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Suicide; Inflammation; Neuroinflammatory Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suicide Attempt Study Group: Adolescents admitted to the Cleveland Clinic inpatient child and adolescent psychiatry unit after suicide attempt. Clinical assessments and blood samples; follow-up for 12 mos.
  Interventions: Other: Clinical assessments and blood samples; follow-up for 12 mos
- Healthy Control Group: Healthy adolescents with no history of suicide attempt. Clinical assessments and blood samples; no 12mo follow-up.
  Interventions: Other: Clinical assessments and blood samples; no 12mo follow-up

INTERVENTIONS:
Other: Clinical assessments and blood samples; follow-up for 12 mos — Kiddie-Sads Present and Lifetime Version Diagnostic Interview, Columbia-Suicide Severity Rating Scale, Suicidal Ideation Questionnaire, Children's Depression Rating Scale-Revised, Multidimensional Anxiety Scale for Children (2nd Ed), Adverse Childhood Experiences Questionnaire, Life Events Checklist-5, Pubertal Development Scale. All assessments administered at baseline, and a smaller subset of assessments administered at discharge and other time points throughout 12 months follow-up. Blood samples taken at baseline (admission to unit) and day of discharge.
  Groups: Suicide Attempt Study Group
Other: Clinical assessments and blood samples; no 12mo follow-up — Kiddie-Sads Present and Lifetime Version Diagnostic Interview, Columbia-Suicide Severity Rating Scale, Suicidal Ideation Questionnaire, Children's Depression Rating Scale-Revised, Multidimensional Anxiety Scale for Children (2nd Ed), Adverse Childhood Experiences Questionnaire, Life Events Checklist-5, Pubertal Development Scale. All assessments administered at baseline, and a smaller subset of assessments administered at discharge time point (5-7 days after baseline). Blood samples taken at baseline and discharge time points (5-7 days after baseline).
  Groups: Healthy Control Group

SUMMARY:
Suicide is one of the most devastating events in society at all levels. The primary goal of this study is to predict suicide in adolescents at risk. We will utilize blood biomarker measurement and clinical risk factor scales to develop a tool to identify adolescents at risk for suicide earlier, which will allow clinicians to prescribe timely treatment and prevent suicide.

DETAILED DESCRIPTION:
Suicide, the second leading cause of death in adolescents (15-24 year olds), is the most tragic complication of a psychiatric condition in this age group. Every year, approximately 157,000 youth receive medical care for suicide related injuries at emergency departments throughout the U.S. Despite some progress, suicide prevention continues to be a daunting task. In adolescents, the risk of a second suicide attempt is approximately 30% after discharge from an inpatient psychiatric unit. Up to 80% of suicidal patients who subsequently died by suicide deny suicidal ideation in their last communication with a health care provider. Therefore, there is an urgent need for the development of biomarkers that can objectively identify which youth are most likely to engage in subsequent suicide attempts.

Several lines of evidence (postmortem studies, genetic studies, biomarker studies) as well as preliminary studies conducted by our group have pointed to neuroinflammation as one of the neurobiological findings observed in suicidal behavior. In particular, the principal investigator and co- investigators have identified S100B - an astrocytic protein, which is a marker of blood brain barrier (BBB) impairment, as a novel biomarker associated with suicidality in adolescents. We are now also investigating three additional and important markers Kynurenic Acid (KYNA), Quinolinic Acid (QUIN), and Picolinic Acid (PIC) identified by Dr. Lena Brundin (Van Andel Institute) to be altered in patients after a suicide attempt. Other studies have reported several other peripheral inflammatory markers (PlMs) including interleukin-1 beta (IL-1ß), interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-α) as associated with suicidality. Hence, PlMs either on their own or along with clinical markers may be particularly useful in predicting future suicide attempts. This study will investigate whether PIM levels, with or without clinical predictors, can be useful at the time of discharge from an inpatient psychiatric unit to predict suicidality in adolescent patients in the subsequent 12 months. The first aim of this study is to determine whether plasma levels of S100B, IL-1ß, IL-6, TNF-α, KYNA, QUIN, and PIC correlate with suicidal behavior (SB). Secondly, this study will investigate if any of the PlMs can predict suicidal attempts. Finally, we will test which combination of clinical risk factors and PlMs is able to most efficiently predict SB post-discharge from the inpatient unit.

Innovative aspects of this study include: 1) The first study to longitudinally investigate levels of PlMs at the time of admission and their change at the time of discharge in adolescent patients being admitted for SB. 2) The first study to investigate whether level of PIMS (alone or in combination with clinical risk factors) at the time of discharge can predict readmissions for SB in the next 12 months. 3) Beside the well-studied PIMs in adult samples, specifically investigate novel biomarkers of inflammation- S100B and 3 markers of the Kynurenine pathway (KYNA, QUIN and PIC).

ELIGIBILITY:
Inclusion Criteria:

Suicide Attempt Study Group:

* 12-18 years of age
* admitted to the Cleveland Clinic inpatient child and adolescent psychiatry unit after suicidal ideations or a suicide attempt

Healthy Control Group:

* 12-18 years of age
* No history of suicide attempt

Exclusion Criteria:

Suicide Attempt Study Group:

* History of autism spectrum disorder
* Non-verbal
* Moderate or severe intellectual disability (IQ<70 and patients in special education full-time)
* Schizophrenia or schizoaffective disorder diagnosis
* Current diagnosis of anorexia or bulimia
* History of generalized tonic-clonic epileptic seizures in last 3 months (If patient does not have a history of seizures, and generalized tonic-clonic seizure was clinically determined to be caused by patient's recent overdose attempt, patient can still be recruited for study if 24 hours has passed since last seizure)
* History of traumatic brain injury, brain tumor, or any major neurological disorder
* Delirium or mood disorder secondary to general medical condition
* Current infection, fever, antibiotic use in the last 2 weeks
* History of autoimmune or immunodeficiency diseases
* Current untreated major endocrine disorder
* Current pregnancy or delivery within the last month
* Diagnosed malnutrition
* Positive urine toxicology for benzodiazepines or opiates on admission
* Current substance use disorder diagnosis and referral for CD assessment upon discharge
* Current diagnosis of morbid obesity or a current BMI greater than 40 kg/m2
* Abnormal complete blood count (CBC)

Healthy Control Group:

* History of any psychiatric diagnosis / treatment (behavioral diagnoses [ADD/ADHD/etc] are okay)
* History of suicidal ideation, behavior, or attempt
* Family history of suicide attempts
* Diagnosis of schizophrenia or bipolar disorder in parents or siblings
* History of autism spectrum disorder
* Moderate or severe intellectual disability (IQ<70 and patients in special education full-time)
* History of generalized tonic-clonic epileptic seizures in last 3 months
* History of headaches or migraines in the last month
* History of traumatic brain injury, brain tumor, or any major neurological disorder
* Delirium or mood disorder secondary to general medical condition
* Current infection, fever, antibiotic use in the last 2 weeks
* History of autoimmune or immunodeficiency diseases
* Current untreated major endocrine disorder
* Current pregnancy or delivery within the last month
* Diagnosed malnutrition
* Report of any substance use in week prior

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The suicide attempt study group will be recruited from all patients (ages 12-18 years) admitted to the Cleveland Clinic inpatient child and adolescent psychiatry unit after a suicide attempt. Healthy adolescent control group (ages 12-18 years) will be recruited through the Cleveland Clinic pediatric outpatient offices.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Relation between levels of peripheral inflammatory markers and suicide attempt | baseline
  Comparison of the levels of peripheral inflammatory markers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) between participants with and without suicide attempt
Relation between levels of peripheral inflammatory markers and suicide attempt | on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Comparison of the levels of peripheral inflammatory markers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) between participants with and without suicide attempt

SECONDARY OUTCOMES:
Change from baseline in peripheral inflammatory marker levels for healthy control group | baseline and on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Comparison of the levels of peripheral inflammatory markers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) between baseline and discharge time points
Change from baseline in peripheral inflammatory marker levels for suicide attempt study group | baseline and on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Comparison of the levels of peripheral inflammatory markers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) between baseline and discharge time points
Relation between levels of peripheral inflammatory markers and Columbia Suicide Severity Rating Scale scores | on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Studying relation between inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) and suicide ideation intensity (scores on Columbia Suicide Severity Rating Scale)
Relation between levels of peripheral inflammatory markers and Suicidal Ideation Questionnaire scores | on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Studying relation between inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) and suicide ideation intensity (Suicidal Ideation Questionnaire)
Relation between levels of peripheral inflammatory markers and depression | on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Studying relation between inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) and depression (scores on Children's Depression Rating Scale, Revised)
Relation between levels of peripheral inflammatory markers and anxiety | on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Studying relation between inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) and anxiety (scores on Multidimensional Anxiety Scale for Children, 2nd Ed)
Relation between levels of peripheral inflammatory markers and trauma | on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Studying relation between inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) and trauma (scores on Adverse Childhood Experiences Questionnaire (ACE) and Life Events Checklist-5 (LEC-5))
Changes in peripheral inflammatory marker levels predicting changes in Columbia Suicide Severity Rating Scale scores | baseline and on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Peripheral inflammatory markers: S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid
Changes in peripheral inflammatory marker levels predicting changes in Suicidal Ideation Questionnaire scores | baseline and on the date of discharge from hospital inpatient unit (average length of admission = 5 days)
  Peripheral inflammatory markers: S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid
Peripheral inflammatory markers as a risk factor for suicide attempts | up to 12 months post-discharge
  Studying inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide attempt risk factors (frequency of attempts)
Peripheral inflammatory markers as a risk factor for suicide ideation intensity (scores on Columbia Suicide Severity Rating Scale) | up to 12 months post-discharge
  Studying inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide ideation intensity risk factors (scores on Columbia Suicide Severity Rating Scale)
Peripheral inflammatory markers as a risk factor for suicide ideation intensity (scores on Suicidal Ideation Questionnaire) | up to 12 months post-discharge
  Studying inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide ideation intensity risk factors (scores on Suicidal Ideation Questionnaire)
Peripheral inflammatory markers as a risk factor for suicide attempt re-admission | up to 12 months post-discharge
  Studying inflammatory biomarkers (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide attempt re-admission risk factors (frequency of re-admissions)
Change in peripheral inflammatory marker levels from baseline to discharge as a risk factor for suicide attempts | up to 12 months post-discharge
  Studying the change in inflammatory biomarkers from baseline to discharge (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide attempt risk factors (frequency of attempts)
Change in peripheral inflammatory marker levels from baseline to discharge as a risk factor for suicide ideation intensity (scores on Columbia Suicide Severity Rating Scale) | up to 12 months post-discharge
  Studying the change in inflammatory biomarkers from baseline to discharge (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide ideation intensity risk factors (scores on Columbia Suicide Severity Rating Scale)
Change in peripheral inflammatory marker levels from baseline to discharge as a risk factor for suicide ideation intensity (scores on Suicidal Ideation Questionnaire) | up to 12 months post-discharge
  Studying the change in inflammatory biomarkers from baseline to discharge (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide ideation intensity risk factors (scores on Suicidal Ideation Questionnaire)
Change in peripheral inflammatory marker levels from baseline to discharge as a risk factor for suicide attempt re-admission | up to 12 months post-discharge
  Studying the change in inflammatory biomarkers from baseline to discharge (S100B, IL-6, IL-1β, TNF-α, kynurenic acid, quinolinic acid, and picolinic acid) as suicide attempt re-admission risk factors (frequency of re-admissions)
Clinical assessment values that predict suicide attempts | up to 12 months post-discharge
  Studying which clinical assessments can help predict suicide attempt (frequency of attempts)
Clinical assessment values that predict suicide ideation intensity scores on Columbia Suicide Severity Rating Scale | up to 12 months post-discharge
  Studying which clinical assessments can help predict suicide ideation intensity scores on Columbia Suicide Severity Rating Scale
Clinical assessment values that predict suicide ideation intensity scores on Suicidal Ideation Questionnaire | up to 12 months post-discharge
  Studying which clinical assessments can help predict suicide ideation intensity scores on Suicidal Ideation Questionnaire
Clinical assessment values that predict suicide attempt re-admission | up to 12 months post-discharge
  Studying which clinical assessments can help predict suicide attempt re-admission (frequency of re-admissions)
Peripheral inflammatory markers in combination with clinical assessments as predictors for suicide attempts | up to 12 months post-discharge
  Studying which combination of inflammatory biomarkers and clinical predictors best predicts future suicide attempts (frequency of attempts)
Peripheral inflammatory markers in combination with clinical assessments as predictors for suicide ideation intensity scores on Columbia Suicide Severity Rating Scale | up to 12 months post-discharge
  Studying which combination of inflammatory biomarkers and clinical predictors best predicts suicide ideation intensity scores on Columbia Suicide Severity Rating Scale
Peripheral inflammatory markers in combination with clinical assessments as predictors for suicide ideation intensity scores on Suicidal Ideation Questionnaire | up to 12 months post-discharge
  Studying which combination of inflammatory biomarkers and clinical predictors best predicts suicide ideation intensity scores on Suicidal Ideation Questionnaire
Peripheral inflammatory markers in combination with clinical assessments as predictors for suicide attempt re-admission | up to 12 months post-discharge
  Studying which combination of inflammatory biomarkers and clinical predictors best predicts future suicide attempt re-admissions (frequency of re-admissions)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Falcone, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No